CLINICAL TRIAL: NCT04825080
Title: Natural History of Asymptomatic Carotid Artery Stenosis in the Modern Era
Brief Title: Carotid Asymptomatic Stenosis
Acronym: CARAS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Rodolfo Pini, MD, PhD, University of Bologna
Other Study IDs: STECA
Record Dates: First submitted 2021-03-26; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Asymptomatic Carotid Artery Stenosis
MeSH Terms: interventions — Ultrasonography, Doppler, Duplex; Computed Tomography Angiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: duplex ultrasound and computed tomography angiography — Identification of carotid artery stenosis > 60% NASCET criteria

SUMMARY:
There is debate on the natural history of asymptomatic severe carotid artery stenosis. Previous studies conducted more than 20 years ago revealed the benefit of carotid endarterectomy compared with medical therapy only on the stroke prevention. However, today it seems that the current medical regimen can reduce the cerebral ischemic event rate in patients with asymptomatic severe carotid artery stenosis to less than 1% per year, making it questionable to choose the surgical treatment.

DETAILED DESCRIPTION:
The Primary end point is to evaluate the rate of cerebral ischemic events (stroke or transient ischemic attack) in patients with asymptomatic carotid artery stenosis > 60% (Nascet criteria) in a 5-year follow-up period. It is a prospective observational study conducted on patients enrolled from January 2019 to March 2020 and with the end of follow-up scheduled in 2025.

The medical therapy recommended includes antihypertensive drugs to maintain good blood pressure control, statin therapy and antiplatelet administration.

Secondary end points are the evaluation of plaque progression, the identification of comorbidities or plaque characteristics associated with a higher risk for cerebral ischemic events and the patient adherence to the best medical therapy in a real world scenario. The global survival and the factors influencing survival will be investigated as well.

Separate analyses are performed for patients with total carotid occlusion or carotid artery re-stenosis.

Patient's cohort: with the hypothesis of 3 neurologic (transient ischemic attack or stroke) events per 100 patients/year during a 5 years follow-up period and consequently a number of 40-50 events (primary outcome), the study cohort with a native asymptomatic carotid artery stenosis will include at least 300 patients. Patients with carotid occlusion or restenosis are evaluated separately for a secondary analysis only.

Patients are prospectively identified and enrolled in a single center vascular surgery ambulatory and a duplex ultrasonography (DUS) laboratory. Carotid artery stenosis are identified and the degree of stenosis >60% (NASCET criteria) is evaluated according to the current guidelines for stenosis identification through blood flow velocities. Patients enrollment goes from January 2019 to March 2020. The investigators prospectively complete the dedicated database including clinical characteristics, cardiovascular risk factors, medical therapy in use, features of the carotid plaque and contralateral carotid status.

Clinical characteristics included in the database: age, sex, hypertension (systolic blood pressure ≥140 or/and diastolic ≥90 mmHg, or specific therapy), dyslipidemia (total cholesterol ≥200 mg/dl or low density lipoprotein ≥120 mg/dl or specific therapy), diabetes mellitus (pre-diagnosed, in therapy with oral hypoglycemic drugs or insulin), current smoking, coronary artery disease (defined as a history of angina pectoris, myocardial infarction or coronary revascularization), chronic obstructive pulmonary disease (defined as chronic bronchitis or emphysema), chronic kidney disease (glomerular filtration rate <60 ml/min), contralateral carotid occlusion, stenosis and atrial fibrillation (paroxysmal or permanent).

Medical therapy: antiplatelet types, anticoagulant therapy, statin therapy, anti hypertensive medical therapy.

Carotid plaque characteristics for the analysis: degree of stenosis (flow measurement analysis), plaque ulcerations and echoluncency.

The follow-up consists of a telephone interview any six months and an annual clinical and duplex examination until a 5-years follow-up is reached or the patient withdraws from the study.

Patients that will be enrolled will sign specific consents. Sensitive patient information will not be available during data analysis. The clinical study will be carried out according to the ethical principles of the Declaration of Helsinki and following the active regulations on observational studies.

Patients who underwent a transient ischemic attach or a stroke within the 6-months before the enrollment are excluded from the study. Any neurological symptom occurred during the follow-up needs to be certified by an in hospital neurologist physical examination.

Statistical analysis: Continuous variables were described with mean and standard deviation. Continuous variables were compared by unpaired Student' t test in case of normal distribution, otherwise by Mann-Whitney's test. The differences between percentages were assessed using Fisher's test or Chi-square test, when appropriate. Univariate analysis will be performed by Kaplan Meier analysis (log-rank test) and single factor Cox analysis . Multivariate analyses with Cox analysis will be performed including factors considered statistical significant (P value ≤ .05) at the univariate analyses. Risk factors were reported as hazard ratio (HR) and 95% of confidence interval (CI). A value of p ≤ .05 (two-tailed) was considered to be significant. The statistical tests were performed using SPSS® 21.0 for Windows® (SPSS, Chicago, Il, USA).

ELIGIBILITY:
Inclusion Criteria:

- asymptomatic carotid artery stenosis (according to the ESVS guidelines) >60% (NASCET criteria) with a physical examination and a DUS at the S. Orsola Malpighi hospital from 2019 to 2025.

Exclusion Criteria:

* Patients submitted to carotid revascularization will be included until the revascularization.
* Patients who underwent a transient ischemic attach or a stroke within the 6-months before the enrollment are excluded from the study
* Restenosis
* Carotid total occlusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are prospectively identified and enrolled in a single center vascular surgery ambulatory and a duplex ultrasonography (DUS) laboratory. Carotid artery stenosis are identified and the degree of stenosis >60% is evaluated according to the current guidelines for stenosis identification through blood flow velocities. Patients enrollment goes from January 2019 to March 2020. The investigators prospectively complete the dedicated database including clinical characteristics, cardiovascular risk factors, medical therapy in use, features of the carotid plaque and contralateral carotid status.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Cerebral ischemic events | 5 years
  Stroke and transient cerebral ischemic events or amaurosis fugax, evaluated by clinical neurologist by clinical examination (National Institutes of Health Stroke Scale, NIHSS or modified Rankin scale, mRS)
Ipsilateral cerebral ischemic events | 5 years
  Ipsilateral stroke and transient cerebral ischemic events or amaurosis fugax, evaluated by clinical neurologist by clinical examination (National Institutes of Health Stroke Scale, NIHSS or modified Rankin scale, mRS)

SECONDARY OUTCOMES:
Plaque progression | 5 years
  Increasing of carotid stenosis from 60%-79% to >80% according with duplex ultrasound flow measurement (Nascent criteria)
Patient's adherence to the medical therapy | 5 years
  adherence to medical drugs prescribed
Survival | 5 years
  Survival rate

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico S. Orsola Malpighi, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No